CLINICAL TRIAL: NCT01663545
Title: Positron Emission Tomography Measurement of Neuroinflammation in Focal Epilepsy
Brief Title: Brain P-gp and Inflammation in People With Epilepsy
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120182; 12-N-0182
Record Dates: First submitted 2012-08-08; First posted 2012-08-13 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2017-10-04

CONDITIONS: Epilepsies, Partial
Keywords: Epilepsy; Epileptic Focus; Inflammation; P-Glycoprotein; PET Imaging
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

* The brain is protected by a barrier that keeps toxins in the blood from reaching the brain. However, this barrier can also keep useful medications from reaching the brain. P-glycoprotein (P-gp) is a brain protein that is part of the blood-brain barrier. The level of P-gp is higher in people with epilepsy than in people without epilepsy. These different levels of P-gp may explain why some people have seizures that do not respond well to medications. Researchers want to see if P-gp can affect the response to epilepsy medications.
* Epilepsy may also be associated with brain inflammation. Researchers also want to look at the part of the brain affected by epilepsy to see if inflammation is present.

Objectives:

* To see if P-gp can affect the response to epilepsy medications.
* To see if inflammation is present in the part of the brain affected by epilepsy.

Eligibility:

* <TAB>Individuals between 18 and 60 years of age who have temporal lobe epilepsy. We plan to study some patients whose seizures are well controlled by drugs, and some whose seizures are not controlled.
* <TAB>
* Healthy volunteers between 18 and 60 years of age.

Design:

* This study requires four or five visits to the NIH Clinical Center over the course of a year. The visits will be outpatient visits and will last from 2 to 5 hours.
* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected.
* All participants will have two positron emission tomography (PET) scans. The scans will take place during different visits. Different drugs will be used in each scan. One drug will be used to temporarily block the effect of P-gp in the brain. The other drug will show areas of inflammation in the brain.
* Participants with epilepsy will have a third PET scan. This scan will also look at P-gp activity in the brain. However, it will not use the drug that blocks the effect of P-gp.
* All participants will also have one magnetic resonance imaging scan. This scan will help show brain function.

DETAILED DESCRIPTION:
Objectives:

1. To study the role of inflammation in focal epilepsy
2. To characterize the BBB state in patients with focal epilepsy using MRI, and compare the results with PET imaging of inflammation
3. To study test-retest replicability of [11C]PBR28 PET scanning.

Study population:

50 participants with drug-resistant focal epilepsy, 25 participants with drug-responsive focal epilepsy and 25 healthy volunteers.

Design:

Screening of enrolled participants will include a medical history, physical exam, and blood and urine laboratory testing. Blood samples will also be used for genetic polymorphism study. Healthy volunteers will receive one or two brain positron emission tomography (PET) scans with [11C]PBR28. Epilepsy participants will receive one or two PET scans with [11C]PBR28). Everyone will receive a brain magnetic resonance imaging (MRI). Some participants will also have a second MRI with gadolinium infusion to measure blood-brain barrier permeability.

Outcome measures:

The primary outcome measure will be the amount of differential [11C]PBR28 uptake between the epileptic focus and the homologous contralateral region. [11C]PBR28 distribution volume (VT) will be measured using an arterial input function. We want to quantify the tracer VT in regions of the brain distant from the epileptic focus, which may be affected by the disease.

We hypothesize that focal epilepsy will be associated with brain inflammation and, therefore, that [11C]PBR28 uptake in the affected side of the brain will be higher than in the contralateral side.

We will study the polymorphism of the translocator protein (TSPO), because TSPO polymorphism has an influence on [11C]PBR28 binding. This polymorphism is due to the non-conservative amino-acid substitution at position 147 from alanine to threonine (Ala147Thr) in the fifth transmembrane domain of the TSPO protein.

ELIGIBILITY:
* INCLUSION CRITERIA:

For patients

* Age 18-60
* Able to give written informed consent.
* Drug resistant participants will be defined as having clinically documented partial seizures with consistent EEG evidence as defined by the 2010 Revised terminology and concepts for organization of seizures and epilepsies and refractory to standard antiepileptic treatment for at least one year prior to enrolling in this study. This criterion will be established by preliminary screening in the NINDS Clinical Epilepsy Section outpatient clinic under protocol 01-N-0139, and if necessary, inpatient video-EEG monitoring. Seizure focus localization will be determined by standard clinical, neurophysiologic, and imaging studies.
* Drug-responsive participants will be defined as having clinically documented partial seizures with consistent EEG evidence as defined by the 2010 Revised terminology and concepts for organization of seizures and epilepsies, seizure-free on standard antiepileptic treatment for at least three months prior to enrolling in this study. This criterion will be established by preliminary screening in the NINDS Clinical Epilepsy Section outpatient clinic under protocol 01-N-0139, and if necessary, inpatient video-EEG monitoring. Seizure focus localization will be determined by standard clinical, neurophysiologic, and imaging studies.
* No prior diagnosis of drug or alcohol abuse or dependence.

For healthy volunteers

* Age 18-60.
* Able to give written informed consent.
* No prior diagnosis of drug or alcohol abuse or dependence.

EXCLUSION CRITERIA:

For patients

* Previous research radiation exposure (X-rays, PET scans etc.) that, together with study procedures, would exceed the NIH RSC 5 rad per year research limit.
* Claustrophobia to a degree that the subject would feel uncomfortable in the MRI machine.
* History of brain disease other than epilepsy.
* Cannot lie on their back for at least two hours.
* Serious medical illness, other than epilepsy.
* Clinically significant laboratory abnormalities.
* Brain abnormality such as a brain tumor, infection, stroke, brain damage from head trauma or blood vessel abnormalities, on an MRI scan.
* Pregnancy or breast feeding.
* Able to get pregnant but does not use birth control.
* Risk for MRI scan, such as a pacemaker or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pump, or shrapnel fragments. Welders and metal workers are also at risk for injury because of possible small metal fragments in the eye of which they may be unaware.
* PBR28 non-binders.
* For drug-responsive subjects: occurrence of a seizure within the last three months.
* NIH employee or staff member

For healthy volunteers

* Clinically significant laboratory abnormalities.
* Unable to have a MRI scan.
* History of neurologic illness or injury with the potential to affect study data interpretation.
* History of seizures, other than in childhood and related to fever.
* Previous research radiation exposure (X-rays, PET scans etc.) that, together with study procedures, would exceed the NIH RSC 5 rad per year research limit.
* Inability to lie flat on camera bed for at least two hours.
* PBR28 non-binders
* Pregnancy or breast feeding.
* Able to get pregnant but does not use birth control.
* NIH employee or staff member

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2012-07-31; Study Completion 2017-10-04

PRIMARY OUTCOMES:
Amount of differential [11C]dLop and [11C]PBR28 uptake between the epileptic focus and the homologous contralateral region | study completion

SECONDARY OUTCOMES:
Secondary Outcome Measure: A secondary goal is to determine if inhibiting P-gp with tariquidar results in increased concentrations of anti-epileptic medications into the CSF, as a surrogate marker for increased penetration of these medication... | study completion

CONTACTS AND LOCATIONS:
Overall Officials: William H Theodore, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Aronica E, Gorter JA, Redeker S, van Vliet EA, Ramkema M, Scheffer GL, Scheper RJ, van der Valk P, Leenstra S, Baayen JC, Spliet WG, Troost D. Localization of breast cancer resistance protein (BCRP) in microvessel endothelium of human control and epileptic brain. Epilepsia. 2005 Jun;46(6):849-57. doi: 10.1111/j.1528-1167.2005.66604.x. PMID 15946326
- [Background] Aronica E, Boer K, van Vliet EA, Redeker S, Baayen JC, Spliet WG, van Rijen PC, Troost D, da Silva FH, Wadman WJ, Gorter JA. Complement activation in experimental and human temporal lobe epilepsy. Neurobiol Dis. 2007 Jun;26(3):497-511. doi: 10.1016/j.nbd.2007.01.015. Epub 2007 Feb 20. PMID 17412602
- [Background] Boer K, Troost D, Spliet WG, van Rijen PC, Gorter JA, Aronica E. Cellular distribution of vascular endothelial growth factor A (VEGFA) and B (VEGFB) and VEGF receptors 1 and 2 in focal cortical dysplasia type IIB. Acta Neuropathol. 2008 Jun;115(6):683-96. doi: 10.1007/s00401-008-0354-6. Epub 2008 Mar 4. PMID 18317782